CLINICAL TRIAL: NCT05779709
Title: The Effectiveness of Reformer Pilates Exercises on Symptoms and Quality of Life in Children With Bladder and Bowel Dysfunction
Brief Title: Reformer Pilates Exerises in Bladder and Bowel Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Clinical Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021/051
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: BLADDER AND BOWEL DYSFUNCTION
Keywords: Reformer; Pilates; Urotherapy; Quality of life; Bladder and bowel dysfunction
MeSH Terms: conditions — Intestinal Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Children between ages 5-18, who were diagnosed with bladder and bowel dysfunction without any neurological abnormalities were invited. Children with neuropathic or anatomical abnormalities in the urinary tract or gastrointestinal tract, inflammatory bowel disease or any other disorder affecting bladder or bowel function and who requested withdrawal from the study at any stage were excluded.
  The children who met the inclusion criteria were invited for pre-intervention meeting and assessments. The aim of study and reformer pilates exercise intervention explained parents and children during the meeting. The children and their parents who want to join exercise sessions during the study were assigned in the reformer pilates group and who did not accept to perform reformer pilates exercises were assigned in the urotherapy group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urotherapy group (Experimental): The purpose of urotherapy education was to teach children to empty the bladder regularly and completely. The standardized urotherapy which included instructions on daily fluid intake of at least 1,200 ml evenly distributed daily as described and voiding at 2-hour intervals until bedtime in which the voiding and defecation positions were taught not to perform avoidance maneuvers. In this training, families were given basic information about the anatomy and physiology of the lower urinary tract (LUT) and anorectum, normal voiding and defecation, fluid consumption and voiding habits of children. The children were allowed to pee whenever they wanted occasionally at any time. Children were also asked to report the number of wet days during 8 weeks
  Interventions: Other: Urotherapy
- Reformer pilates group (Experimental): The basic pilates principles were explained to the children. The diaphragmatic breathing, neutral position of the pelvis, centering and pelvic floor control were teached with appropriate language for their age. Verbal help were given to maintain centering during each movement. The exercises (30 min) were started by doing 10 repetitions in combination with diaphragm breathing, and progressed 12 repetitions after 3 weeks, 15 repetitions after 6 weeks (frog series, leg circles series, hundred series, box series, side splits series).İndividual reformer pilates training consisting of 30 minutes two days a week was given to the exercise group by an expert physiotherapist for 8 weeks.
  Interventions: Other: exercise; Other: Urotherapy

INTERVENTIONS:
Other: exercise — Reformer pilates is a specific type that provides resistance exercise at certain weights with the pulley system relying basically on the same principles. Pilates exercises provide breathing and activation of the deep stabilizing muscles of the trunk in coordination with the PFMs. It includes exercises that focus on pelvic stability, mobility and body alignment. PFMs activation is carried out simultaneously with the trunk muscles in various positions in coordination with breathing.
  Arms: Reformer pilates group
Other: Urotherapy — Urotherapy includes education of the child and family, diet (adequate fiber and fluid consumption), regular optimal voiding, daily physical activity, teaching normal toilet use, pelvic floor muscle training and relaxation

SUMMARY:
Bladder and bowel dysfunction (BBD) describes the urinary tract symptoms associated with bowel complaints. Urotherapy and pharmacological treatments are used in conservative BBD treatment. Pilates is an exercise method that includes a series of movements that both strengthen and increase flexibility of the entire body without focusing on a specific muscle. Reformer pilates is a specific type that provides resistance exercise at certain weights with the pulley system relying basically on the same principles. Pilates exercises provide breathing and activation of the deep stabilizing muscles of the trunk in coordination with the pelvic floor muscles (PFMs).

Despite the increasing number of health care professionals using the pilates-based approach in rehabilitation. The pilates-based exercises in rehabilitation is still insufficient in the literature7. To our knowledge, none of studies which were investigated the usefulness of pilates-based exercise principle in children with BBD. This study was aimed to investigate the effect of reformer pilates exercises on bladder and bowel dysfunction symptoms and quality of life in children with bladder and bowel dysfunction.

DETAILED DESCRIPTION:
Bladder and bowel dysfunction (BBD) describes the urinary tract symptoms associated with bowel complaints. BBD symptoms are thought to represent 40% of pediatric urology consultations. In children who do not have any neurological or physiological problems, micturition and defecation occur with the coordinated work of the involuntary bladder and bowel, voluntary contracting external urethral sphincter and external anorectal sphincter. For normal micturition and defecation, the pelvic floor muscles must be able to relax properly. This relaxation may not be achieved even in children with no neurological or physiological problems.

Urotherapy and pharmacological treatments are used in conservative BBD treatment. Urotherapy includes education of the child and family, diet (adequate fiber and fluid consumption), regular optimal voiding, daily physical activity, teaching normal toilet use, pelvic floor muscle training and relaxation. Pilates is an exercise method that includes a series of movements that both strengthen and increase flexibility of the entire body without focusing on a specific muscle. It includes exercises that can work the pelvic floor muscles (PFMs), while avoiding intense abdominal contractions, holding breath, or straining that can create increased pressure on the pelvic floor.

Reformer pilates is a specific type that provides resistance exercise at certain weights with the pulley system relying basically on the same principles. Pilates exercises provide breathing and activation of the deep stabilizing muscles of the trunk in coordination with the PFMs. It includes exercises that focus on pelvic stability, mobility and body alignment. PFMs activation is carried out simultaneously with the trunk muscles in various positions in coordination with breathing. Such exercises are known to have an important role related to continence, maintenance of intra-abdominal pressure and respiratory mechanics.

Despite the increasing number of health care professionals using the pilates-based approach in rehabilitation. The pilates-based exercises in rehabilitation is still insufficient in the literature. To our knowledge, none of studies which were investigated the usefulness of pilates-based exercise principle in children with BBD. This study was aimed to investigate the effect of reformer pilates exercises on bladder and bowel dysfunction symptoms and quality of life in children with bladder and bowel dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Children between ages 5-18,
* Diagnosed with bladder and bowel dysfunction without any neurological abnormalities

Exclusion Criteria:

* Children with neuropathic or anatomical abnormalities in the urinary tract or gastrointestinal tract, inflammatory bowel disease or any other disorder affecting bladder or bowel function and who requested withdrawal from the study at any stage were excluded.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Voiding Disorders Symptom Scoring | 8 weeks
  Voiding disorders symptom scoring was developed by Akbal et al. First, it was formed as an empirical questionnaire consisting of questions about day/night symptoms, micturition, defecation habits and quality of life. Then Akbal et al. excluded the question about quality of life and achieved a 90% rate in the specificity and sensitivity study they conducted for 8.5 points and above. The questionnaire includes 13 questions for symptoms and 1 question for quality of life. The maximum score is 35, the minimum score is 0.
Bladder and Bowel Dysfunction Questionnaire | 8 weeks
  The Bladder and Bowel Dysfunction Questionnaire (BBDQ) was used to assess bowel and bladder dysfunctions. Drzewiecki et al. found that this questionnaire was reliable in detecting and evaluating the non-neuropathic pediatric BBDQ. The questionnaire has 14-item and scores for all questions except the first question range from 0 to 4 points, with 0 points indicating no complaints and 4 points indicating the most severe complaints. In the first validation study performed on this questionnaire, 11 points or 52 points were shown as the threshold for BBDQ.
Pediatric İncontinence Questionnaire | 8 weeks
  Bower et al. developed the Pediatric İncontinence Questionnaire (PinQ), a cross-cultural tool specific to children with lower urinary tract dysfunction. This instrument has proven to be a reliable and valid tool for measuring the holistic impact of bladder dysfunction in children, and has been recommended for assessing the quality of life in children with urinary incontinence. The questionnaire was also used to measure changes in quality of life during therapy. The PinQ consists of 20 items. Items have five response options following the Likert scale: 0 no, 1 difficult, 2 sometimes, 3 often, and 4 always. The maximum total score is 80 and higher score means a lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Yakut, Study Chair — Hasan Kalyoncu University
Locations (1):
- Hasan kalyoncu üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguiar LM, Franco I. Bladder Bowel Dysfunction. Urol Clin North Am. 2018 Nov;45(4):633-640. doi: 10.1016/j.ucl.2018.06.010. Epub 2018 Sep 7. PMID 30316317
- [Background] Wennergren HM, Oberg BE, Sandstedt P. The importance of leg support for relaxation of the pelvic floor muscles. A surface electromyograph study in healthy girls. Scand J Urol Nephrol. 1991;25(3):205-13. doi: 10.3109/00365599109107948. PMID 1947848
- [Background] Berry A. Helping children with dysfunctional voiding. Urol Nurs. 2005 Jun;25(3):193-200; quiz 201. PMID 16050350
- [Background] Ladi-Seyedian SS, Sharifi-Rad L, Kajbafzadeh AM. Management of Bladder Bowel Dysfunction in Children by Pelvic Floor Interferential Electrical Stimulation and Muscle Exercises: A Randomized Clinical Trial. Urology. 2020 Oct;144:182-187. doi: 10.1016/j.urology.2020.07.015. Epub 2020 Jul 25. PMID 32717244
- [Background] Lausen A, Marsland L, Head S, Jackson J, Lausen B. Modified Pilates as an adjunct to standard physiotherapy care for urinary incontinence: a mixed methods pilot for a randomised controlled trial. BMC Womens Health. 2018 Jan 12;18(1):16. doi: 10.1186/s12905-017-0503-y. PMID 29329567
- [Background] Pedriali FR, Gomes CS, Soares L, Urbano MR, Moreira EC, Averbeck MA, de Almeida SH. Is pilates as effective as conventional pelvic floor muscle exercises in the conservative treatment of post-prostatectomy urinary incontinence? A randomised controlled trial. Neurourol Urodyn. 2016 Jun;35(5):615-21. doi: 10.1002/nau.22761. Epub 2015 Mar 21. PMID 25809925
- [Background] Kaya Narter F, Tarhan F, Narter KF, Sabuncu K, Alay Eser R, Akin Y, Ay P. Reliability and validity of the Bladder and Bowel Dysfunction Questionnaireamong Turkish children. Turk J Med Sci. 2017 Dec 19;47(6):1765-1769. doi: 10.3906/sag-1601-122. PMID 29306236
- [Background] Akbal C, Genc Y, Burgu B, Ozden E, Tekgul S. Dysfunctional voiding and incontinence scoring system: quantitative evaluation of incontinence symptoms in pediatric population. J Urol. 2005 Mar;173(3):969-73. doi: 10.1097/01.ju.0000152183.91888.f6. PMID 15711352
- [Background] Bower WF, Sit FK, Bluyssen N, Wong EM, Yeung CK. PinQ: a valid, reliable and reproducible quality-of-life measure in children with bladder dysfunction. J Pediatr Urol. 2006 Jun;2(3):185-9. doi: 10.1016/j.jpurol.2005.07.004. Epub 2005 Aug 19. PMID 18947606